CLINICAL TRIAL: NCT06733376
Title: Evaluating Evidence Based Options for Initial PTSD Treatment Non-Responders
Brief Title: Evaluating Evidenced Based Options for PTSD Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Philip Held, Research Director, Rush University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23091403
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: ptsd treatment
MeSH Terms: conditions — Combat Disorders | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Initial Course of Cognitive Processing Therapy (Other): All participants will start in Arm 1 where they receive 10-sessions of Cognitive Processing Therapy.
  Interventions: Behavioral: Cognitive Processing Therapy
- Subsequent Treatment (Active Comparator): At one-week follow up after initial Cognitive Processing Therapy, participants whose scores are 28 or above on the PTSD Checklist for DSM-5 will be offered a subsequent course of treatment.
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Prolonged Exposure; Behavioral: Skills Training for Affective and Interpersonal Regulation

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is a first-line intervention for the treatment of PTSD that focuses on changing unhelpful patterns of thinking.
  Other Names: CPT
Behavioral: Prolonged Exposure — Prolonged Exposure is an evidence-based treatment for PTSD that helps to reduce the intensity of distress by gradually exposing participants to trauma-related memories, feelings, and situations in real life.
  Other Names: PE
  Arms: Subsequent Treatment
Behavioral: Skills Training for Affective and Interpersonal Regulation — Skills Training for Affective and Interpersonal Regulation (STAIR) is a evidence-based treatment geared towards helping regulate emotional and interpersonal needs of those with PTSD.
  Other Names: STAIR
  Arms: Subsequent Treatment

SUMMARY:
This study will look at:

How practical it is to offer another round of proven therapy. How effective different therapy options are for people who didn't respond to the first treatment.

The goal is to improve personalized care by:

Identifying factors that might predict how someone will respond to a second treatment.

Creating a simple tool to spot people who might not respond to treatment early, so they can start a different option sooner.

The findings will help improve PTSD care by offering better follow-up treatments and matching patients with the approach that works best for them.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older
* Are fluent in English
* Have experienced a Criterion A traumatic event during their lifetime
* Have a PTSD diagnosis verified via the Clinician Administered PTSD Scale for DSM-5
* Are interested in receiving evidence-based treatment for PTSD and able to attend 10 therapy sessions over the course of 2 weeks (10 days) and could possibly attend another 10 sessions of a subsequent treatment (additional CPT sessions, PE, or STAIR)
* Are willing and able to complete self-report measures and clinician-rated assessments at multiple timepoints over the course of the study

Exclusion Criteria:

* The index traumatic event occurred in the past month
* They are currently suicidal or homicidal (i.e., current plan and imminent intent)
* They have unmanaged psychosis or mania
* They have not been on a stable dose of psychotropic medication for at least one month at the time of the baseline assessment
* They have completed an evidence-based cognitive behavioral PTSD treatment in the past three months or are currently engaged in an evidence-based PTSD treatment (CPT, PE)
* They have an intellectual disability or significant cognitive impairment that would prevent them from engaging in treatment
* They have a serious or unstable medical illness or instability for which hospitalization may be likely within the next year
* They have an active substance use disorder (within the past three months) that would require immediate medical observation if substance was abruptly discontinued
* They are involved with current legal actions related to their index trauma
* They have a visual or auditory impairment that would prevent them from fully participating in study activities
* They, at the time of consent, appear to have extenuating life circumstances (i.e., unstable housing, no internet access, etc.) which, in the judgement of the study team, could affect the ability to deliver interventions with fidelity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline to 6 month follow up
  A self-report measure of PTSD symptom severity
Clinician Administered PTSD Scale for DSM-5 | Baseline to 6 mont follow up
  A clinician-rated assessment of PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No